CLINICAL TRIAL: NCT01660893
Title: A Phase III, Multi-Center, Randomized, Double-Blind, Parallel-Groups Clinical Trial Comparing the Efficacy and Safety of Intranasally Administered Kovacaine Mist to Tetracaine Alone and to Placebo for Anesthetizing Maxillary Teeth in Adults
Brief Title: Comparison of Intranasal Kovacaine Mist, Tetracaine Alone, and Placebo for Anesthetizing Maxillary Teeth
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR 3-01
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Anesthesia
Keywords: operative; dental procedure
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kovacaine Mist, 3 sprays unilateral (Experimental): Tetracaine HCl 3% and oxymetazoline HCl 0.05%
  Interventions: Drug: Tetracaine HCl 3% and oxymetazoline HCl 0.05%
- Tetracaine Only, 3 sprays unilateral (Experimental): Tetracaine HCl 3%
  Interventions: Drug: Tetracaine HCl 3%
- Placebo, 3 sprays unilateral (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetracaine HCl 3% and oxymetazoline HCl 0.05% — 3 unilateral intranasal sprays per dose
  Other Names: Kovacaine Mist
  Arms: Kovacaine Mist, 3 sprays unilateral
Drug: Tetracaine HCl 3% — 3 unilateral intranasal sprays per dose
  Arms: Tetracaine Only, 3 sprays unilateral
Drug: Placebo — 3 unilateral intranasal sprays per dose
  Arms: Placebo, 3 sprays unilateral

SUMMARY:
The purpose of this study is to compare the efficacy of Kovacaine Mist, Tetracaine only, and Placebo for inducing pulpal anesthesia of the maxillary teeth in adults.

DETAILED DESCRIPTION:
The study will employ a multi-center, randomized, double-blind, placebo-controlled, parallel-groups design to assess the safety and efficacy of Kovacaine Mist delivered intranasally for inducing pulpal anesthesia of maxillary teeth numbers 4 to 13 (maxillary right second premolar to maxillary left second premolar) sufficient to allow completion of the Study Dental Procedure.

A total of 140 subjects, randomized 2:2:1 (Kovacaine Mist:Tetracaine alone:Placebo) will be enrolled to achieve 125 completed subjects; a total of 50 Kovacaine Mist subjects, 50 tetracaine alone subjects and 25 placebo subjects. Recruitment will be from diverse dental patient populations. At the two study sites, a balanced enrollment of 70 subjects each is planned to allow for a potential 10% drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Need for an operative restorative dental procedure requiring local anesthesia for a single vital maxillary tooth (other than a maxillary first, second, or third molar) with no evidence of pulpal pathology.
* Normal lip, nose, eyelid, and cheek sensation.
* Able to understand and sign the study informed consent document, communicate with the investigators, and understand and comply with the requirements of the protocol.
* Patency of the naris ipsilateral to the tooth undergoing the Study Dental Procedure.
* Resting heart rate (HR) between 55 and 100 beats per minute (bpm), inclusive.
* Seated systolic blood pressure (SBP) between 95 and 140 mm Hg, inclusive and seated diastolic blood pressure (DBP) between 60 and 90 mm Hg, inclusive.

Exclusion Criteria:

* Inadequately controlled hypertension (blood pressure greater than 140/90 mm Hg).
* Inadequately controlled active thyroid disease of any type.
* Frequent nose bleeds (≥ 5 per month).
* Having received dental care requiring a local anesthetic within the last 24 hours.
* History of allergy to or intolerance of tetracaine, benzyl alcohol, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreen).
* History of allergy or hypersensitivity to articaine, oxymetazoline, epinephrine, or sulfite preservatives.
* Use of a monoamine oxidase inhibitor within the 3 weeks preceding study entry.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females of child-bearing potential will be required to take a urine pregnancy test on the day of, but prior to, study drug administration to rule out pregnancy.)
* Having received any investigational drug and/or participation in any clinical trial within 30 days prior to study participation.
* Having used oxymetazoline or phenylephrine nasal spray, nasal irrigation, or other nasal or oral decongestant on the day of the study procedure.
* History of congenital or idiopathic methemoglobinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Moore, DMD/PhD/MPH, Study Director — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Family and Cosmetic Dentistry, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Started | 10 | 10 | 6
Completed | 10 | 10 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral | Total
Number analyzed (Participants) | 10 | 10 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (10.22) | 33.3 (11.10) | 32.7 (9.85) | 32.4 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 4 | 20
  Male | 2 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 9 | 9 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 8 | 9 | 6 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Completion of the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic (Yes/no).
Time Frame: at 15 minutes with a 3 minute window
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants
  Success | 5 | 2 | 0
  Failure | 5 | 8 | 6

2. Secondary Outcome: Intraoral Soft-tissue Anesthesia (Yes/no)
Description: Number of patients who reported no pain when incisive papilla and greater palatine foramen soft-tissue was tested with a probe
Time Frame: at 15 minutes with a 3 minute window
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants
  Incisive Papilla | 7 | 5 | 2
  Greater Palatine Foramen | 2 | 1 | 1

3. Secondary Outcome: Number of Participants With Heart Rate Higher Than 125 Bpm
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Heart Rate Lower Than 50 Bpm
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With an Increase From Baseline in Systolic Blood Pressure Greater Than or Equal to 25 mm Hg and to a Value Higher Than 160 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With a Decrease From Baseline in Systolic Blood Pressure Greater Than or Equal to 15 mm Hg and to a Value Lower Than 90 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With an Increase From Baseline in Diastolic Blood Pressure Greater Than or Equal to 15 mm Hg and to a Value Higher Than 90 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With a Decrease From Baseline in Diastolic Blood Pressure Greater Than or Equal to 15 mm Hg and to a Value Lower Than 90 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
Participants | 0 | 0 | 0

9. Secondary Outcome: Absolute Maximum Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
mmHg
  Systolic Blood Pressure | 12.8 (6.05) | 3.5 (8.34) | 1.2 (7.25)
  Diastolic Blood Pressure | 11.2 (5.35) | 4.5 (4.12) | 6.2 (8.84)

10. Secondary Outcome: The Profile Over Time of Heart Rate
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
bpm
  Pre-Study | 76.9 (9.07) | 69.1 (7.95) | 81.0 (8.10)
  10 Minutes | 69.6 (8.3) | 67.1 (7.03) | 75.8 (8.61)
  30 Minutes | 64.6 (9.48) | 64.5 (6.36) | NA (NA) — Data was not collected as study dental procedure was still ongoing
  45 Minutes | 69.6 (8.65) | 64.3 (5.70) | 73.8 (8.30)
  60 Minutes | 67.3 (11.34) | 65.3 (8.31) | 70.2 (5.04)
  90 Minutes | 67.1 (7.74) | 64.3 (8.39) | 72.0 (7.56)
  120 Minutes | 68.4 (6.31) | 65.0 (8.43) | 70.8 (7.57)

11. Secondary Outcome: Alcohol Sniff Test
Description: The change from screening in the the distance from the nose (in centimeters) that a patient is able to detect the smell of an alcohol swab.
Time Frame: administered at approximately 24 hours after drug administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
cm | 0.4 (5.44) | 0.8 (7.69) | 2.1 (2.94)

12. Secondary Outcome: The Profile Over Time of Systolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
mmHg
  Pre-Study | 113.0 (8.23) | 116.1 (11.0) | 125.5 (6.19)
  10 Minutes | 116.5 (6.82) | 114.2 (5.51) | 118.8 (8.77)
  30 Minutes | 123.0 (11.34) | 110.0 (4.24) | NA (NA) — Data was not collected as study dental procedure was still ongoing
  45 Minutes | 118.5 (9.26) | 113.6 (9.31) | 118.8 (10.44)
  60 Minutes | 116.1 (9.68) | 113.3 (7.27) | 121.7 (12.39)
  90 Minutes | 117.7 (8.34) | 112.0 (6.93) | 119.7 (8.89)
  120 Minutes | 119.5 (10.89) | 113.7 (9.31) | 119.2 (9.50)

13. Secondary Outcome: The Profile Over Time of Diastolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
mmHg
  Pre-Study | 74.1 (5.09) | 73.0 (7.09) | 77.7 (7.17)
  10 Minutes | 77.9 (7.06) | 73.8 (5.65) | 75.5 (4.23)
  30 Minutes | 81.0 (6.96) | 70.0 (1.41) | NA (NA) — Data was not collected as study dental procedure was still ongoing
  45 Minutes | 76.4 (5.8) | 72.2 (6.03) | 74.2 (7.81)
  60 Minutes | 76.1 (6.62) | 75.9 (6.52) | 77.8 (7.68)
  90 Minutes | 80.5 (8.78) | 73.1 (6.40) | 78.8 (7.28)
  120 Minutes | 79.1 (10.91) | 72.1 (8.13) | 77.7 (8.55)

14. Secondary Outcome: Absolute Maximum Change From Baseline in Heart Rate
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Number analyzed (Participants) | 10 | 10 | 6
bpm | 3.4 (8.62) | 3.5 (7.09) | 2.3 (7.55)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Kovacaine Mist, 3 Sprays Unilateral | Tetracaine Only, 3 Sprays Unilateral | Placebo, 3 Sprays Unilateral
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Mist, 3 Sprays Unilateral (N=10) | Tetracaine Only, 3 Sprays Unilateral (N=10) | Placebo, 3 Sprays Unilateral (N=6)
Oral discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0 — Runny nose
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 — Intranasal stinging or burning
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 — Abnormal taste
Headache (Nervous system disorders) | 1 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 3 | 2 | 0 — Tearing or watery eyes
Vision blurred (Eye disorders) | 2 | 0 | 0
Hypoaesthesia eye (Eye disorders) | 1 | 1 | 0 — Numbness around eye
Ear discomfort (Ear and labyrinth disorders) | 1 | 1 | 0
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Intranasal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Anaesthetic Complication (Injury, poisoning and procedural complications) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No